CLINICAL TRIAL: NCT04195945
Title: Randomized Phase 2 Trial of CPX-351 (Vyxeos) vs. CLAG-M (Cladribine, Cytarabine, G-CSF, and Mitoxantrone) in Medically Less-Fit Adults With Acute Myeloid Leukemia (AML) or Other High-Grade Myeloid Neoplasm
Brief Title: CPX-351 or CLAG-M Regimen for the Treatment of Acute Myeloid Leukemia or Other High-Grade Myeloid Neoplasms in Medically Less-Fit Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1005577; NCI-2019-07640 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10330 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia; Myeloid Neoplasm
Keywords: Myeloid and Monocytic Leukemia; Other Hematopoietic
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Monocytic, Acute | interventions — CPX-351; Injections; Cytarabine; Daunorubicin; Liposomes; Cladribine; 2'-chloro-2'-deoxyadenosine; pegylated granulocyte colony-stimulating factor; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (CPX-351) (Experimental): INDUCTION: Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity. Patients who achieve a response other than an MRDneg CR receive a second course of CPX-351 intravenously IV over 90 minutes on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity.
  POST-REMISSION: Patients who achieve a CR/CRi receive a reduced dose of CPX-351 IV over 90 minutes on days 1, 3, and 5 for up to 4 additional courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Other: Questionnaire Administration; Other: Quality-of-Life Assessment
- Arm II (CLAG-M) (Experimental): INDUCTION: Patients receive cladribine IV over 2 hours on days 1-5, cytarabine IV over 2 hours on days 1-5, G-CSF SC on days 0-5, and mitoxantrone IV over 60 minutes on days 1-3 in the absence of disease progression or unacceptable toxicity. Patients who achieve a response other than an MRDneg CR receive a second course of cladribine IV over 2 hours on days 1-5, cytarabine IV over 2 hours on days 1-5, G-CSF SC on days 0-5, and mitoxantrone IV over 60 minutes on days 1-3 in the absence of disease progression or unacceptable toxicity.
  POST-REMISSION: Patients who achieve a CR/CRi receive an intermediate dose of cytarabine IV over 2 hours on days 1-6 for up to 4 additional courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Biological: Recombinant Granulocyte Colony-Stimulating Factor; Drug: Mitoxantrone; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos; Daunorubicin and Cytarabine (Liposomal)
  Arms: Arm I (CPX-351)
Drug: Cladribine — Given IV
  Other Names: 105014; 105014-F; 2-Chloro-2-Deoxyadenosine; 2-Chlorodeoxyadenosine; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
  Arms: Arm II (CLAG-M)
Drug: Cytarabine — Given IV
  Other Names: ARA-cell; Arabine; Arabinofuranosylcytosine; Aracytidine; Beta-Cytosine Arabinoside; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920
  Arms: Arm II (CLAG-M)
Biological: Recombinant Granulocyte Colony-Stimulating Factor — Given SC
  Other Names: 143011-72-7; Recombinant Colony-Stimulating Factor 3; rhG-CSF
  Arms: Arm II (CLAG-M)
Drug: Mitoxantrone — Given IV
  Other Names: Dihydroxyanthracenedione; Mitozantrone
  Arms: Arm II (CLAG-M)
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies how well CPX-351 or the CLAG-M regimen (consisting of the drugs cladribine, cytarabine, G-CSF, and mitoxantrone) works in treating medically less-fit patients with acute myeloid leukemia or other high-grade myeloid neoplasms. Drugs used in chemotherapy, such as CPX-351, cladribine, cytarabine, G-CSF, and mitoxantrone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving CPX-351 or the CLAG-M regimen at doses typically used for medically-fit patients with acute myeloid leukemia may work better than reduced doses of CPX-351 in treating medically less-fit patients with acute myeloid leukemia or other high-grade myeloid neoplasms.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms in a 1:1 fashion. ARM I = CPX-351; ARM II = CLAG-M.

ARM I (INDUCTION): Patients receive CPX-351 intravenously (IV) over 90 minutes on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity. Patients who achieve a response other than an MRDneg CR receive a second course of CPX-351 intravenously IV over 90 minutes on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity.

ARM I (POST-REMISSION): Patients who achieve a CR or CR with incomplete hematologic recovery (CRi) receive a reduced dose of CPX-351 IV over 90 minutes on days 1, 3, and 5 for up to 4 additional courses in the absence of disease progression or unacceptable toxicity.

ARM II (INDUCTION): Patients receive cladribine IV over 2 hours on days 1-5, cytarabine IV over 2 hours on days 1-5, G-CSF subcutaneously (SC) on days 0-5, and mitoxantrone IV over 60 minutes on days 1-3 in the absence of disease progression or unacceptable toxicity. Patients who achieve a response other than an MRDneg CR receive a second course of cladribine IV over 2 hours on days 1-5, cytarabine IV over 2 hours on days 1-5, G-CSF SC on days 0-5, and mitoxantrone IV over 60 minutes on days 1-3 in the absence of disease progression or unacceptable toxicity.

ARM II (POST-REMISSION): Patients who achieve a CR/CRi receive an intermediate dose of cytarabine IV over 2 hours on days 1-6 for up to 4 additional courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of untreated "high-grade" myeloid neoplasm (>=10% blasts in blood or bone marrow) or AML other than acute promyelocytic leukemia (APL) with t(15;17)(q22;q12) or variants according to the 2016 World Health Organization (WHO) classification. Outside diagnostic material is acceptable to establish diagnosis; submission of peripheral blood specimen for flow cytometry performed at the study institution should be considered. Diagnostic material must have been submitted for cytogenetic and/or molecular testing as clinically appropriate
* Treatment-related mortality (TRM) score >= 13.1 as calculated with simplified model
* The use of hydroxyurea before enrollment is permitted; hydroxyurea should be discontinued prior to start of study treatment. Patients with symptoms/signs of hyperleukocytosis or white blood cells (WBC) > 100,000/uL or with concern for other complications of high tumor burden or leukostasis (e.g. hypoxia, disseminated intravascular coagulation) can be treated with leukapheresis or may receive up to 2 doses of cytarabine (up to 500 mg/m^2) any time prior to enrollment
* Patients may have received low-intensity treatment (e.g. azacitidine/decitabine, lenalidomide, growth factors) for antecedent low-grade myeloid neoplasm (i.e. < 10% blasts in blood and bone marrow)
* Bilirubin < 2.0 mg/mL unless elevation is thought to be due to hepatic infiltration by neoplastic cells, Gilbert's syndrome, or hemolysis (assessed within 14 days prior to study day 0)
* Left ventricular ejection fraction (LVEF) >= 45%, assessed within 12 months prior to registration, e.g. by multigated acquisition scan (MUGA) scan or echocardiography or another appropriate diagnostic modality
* Women of childbearing potential and men must agree to use adequate contraception beginning at the signing of the consent until at least 4 weeks after the last dose of study drug
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Myeloid blast crisis of chronic myeloid leukemia (CML), unless patient is not considered candidate for tyrosine kinase inhibitor treatment
* Concomitant illness associated with a likely survival of < 1 year
* Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with anti-microbials and/or controlled or stable. Patients with fever thought to be likely secondary to leukemia are eligible
* Known hypersensitivity to any study drug used in this trial
* Pregnancy or active breast feeding
* Concurrent treatment with any other approved or investigational anti-leukemia agent. Treatment with a FLT3-inhibitor for FLT3-mutated AML is permissible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
3-month overall survival (OS) | Up to 3 months from date of start of protocol therapy
  Will evaluate whether CPX-351 or cladribine, cytarabine, granulocyte colony-stimulating factor (G-CSF), and mitoxantrone (CLAG-M), at doses typically used for medically-fit adults with AML, improve 3-month overall survival in medically-unfit adults with AML compared to attenuated dose CPX-351 as used in our previous institutional trial (32 units/m2 per dose).

SECONDARY OUTCOMES:
Complete remission (CR) rates | Up to 5 years post treatment
  Will compare CR rates between the study arms.
MRDneg CR rates | Up to 5 years post treatment
  Will compare MRDneg CR rates between the study arms.
Response duration | Up to 5 years post treatment
  Will compare response duration between the study arms.
Relapse-free survival | Up to 5 years post treatment
  Will compare RFS between the study arms.
Incidence of adverse events | Up to 5 years post treatment
  Will use the CTCAE (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events) version 5.0 for toxicity and adverse event reporting. Will describe the toxicity profile and infectious complications of each study treatment.
30-day mortality rate | At 30 days
60-day mortality | At 60 days
Quality of life (QOL): questionnaire | Up to 5 years post treatment
  QOL of patients will be assessed longitudinally using the European Organization for Research and Treatment of Cancer (EORTC) core QOL questionnaire (QLQ-C30) and the newly developed acute myeloid leukemia-specific QOL instrument.
Patient use of medical resources (e.g. transfusions) | Up to 5 years post treatment
  Electronic medical chart review to enumerate the number of platelet and red blood cell transfusions administered, the number of days spent on IV antimicrobial therapy, and the number of days spent in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Roland Walter, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT04195945/ICF_000.pdf